CLINICAL TRIAL: NCT02149251
Title: Does Preimplantation Genetic Diagnosis for Sex Selection Affect the Pregnancy and Miscarriage Rates in Women With an Expected Good Ovarian Response Undergoing IVF/ICSI Cycles?
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Other Study IDs: Gany 125
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy
Keywords: Pre-genetic diagnosis; ICSI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-genetic diagnosis: Women in this group had ICSI and PGD to exclude genetically affected children or for sex selection
  Interventions: Genetic: Pre-genetic diagnosis
- Control group: This group will include women who had IVF without PGD

INTERVENTIONS:
Genetic: Pre-genetic diagnosis
  Groups: Pre-genetic diagnosis

SUMMARY:
Records of women who had Pre-genetic diagnosis (PGD) over the last 3 years will be reviewed and its outcome will be compared to other records of women who had IVF/ICSI without PGD.

DETAILED DESCRIPTION:
Records of women who had PGD over the last 3 years will be reviewed and its outcome will be compared to other records of women who had IVF/ICSI without PGD Before starting the PGD process couples were seen by a geneticist to assess the feasibility of the procedure for each couple. Couples were then counselled by a gynaecologist specialised in IVF to assess their fertility status and explain the whole procedure including the expected success rates and risks of IVF.

Women had standard pituitary down-regulation with GnRHa (Triptorelin 0.1mg, Decapeptyl® Ferring, Germany) day 7 after ovulation of previous cycle or on day 21 of the oral contraceptive cycles. GnRHa was continued for 2 weeks. Human menopausal gonadotrophin(HMG) (Merional ®IBSA) 150-300 IU/day was administered until the day of HCG administration, Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG.

After fertilization, biopsy was obtained from cleavage stage embryos. FISH analysis was used to distinguish embryos with balanced and unbalanced chromosomal abnormalities for carriers of structural chromosomal aberrations. In the analysis of translocations, unique FISH probes that flank the breakpoints of each translocation or that require the use of subtelomeric probes (specific to the chromosome ends of the translocated segments) for each affected individual must be designed and validated to detect normal and balanced products in embryonic tissue.

The principle of PGD by FISH is that target-specific DNA probes labelled with different fluorochromes or haptens can be used to detect the copy number of specific loci, and thereby to detect chromosome imbalance associated with meiotic segregation of chromosome rearrangements which includes the Robertsonian translocations, reciprocal translocations, inversions, and complex rearrangements. FISH can also be used to select female embryos in families with X-linked disease Polymerase chain reaction (PCR) has been used to diagnose monogenic disorders. PCR is used to amplify sufficient DNA from embryo cells . A blastomere is placed in a solution that lyses the cell and releases the DNA and the PCR reaction mix is then added to begin the PCR. Because of its high sensitivity, contamination of the study sample with extraneous DNA is a danger and has led to the adoption of rigorous laboratory procedures and standards, such as the use of intracytoplasmic sperm injection.

PGD analysis results were available on day 5 after oocyte retrieval. If possible, 2 unaffected embryos were transferred and the rest of the unaffected embryos were cryopreserved.

Women were followed up and a pregnancy test was performed to detect pregnancy, pregnant women were followed up and any pregnancy complications were recorded

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI
* Age 20-40 years

Exclusion Criteria:

* Frozen embryos
* Poor responders defined according to the Bologna criteria
* Recurrent miscarriage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women who had IVF/ICSI over the past 3 years in Dar AlTeb subfertility centre will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 11006 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Miscarriage | 28 weeks after the pregnancy test

SECONDARY OUTCOMES:
pregnancy | 5 weeks after embryo transfer
  pregnancy was defined as the presence of an intrauterine gestational sac 5 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (1):
- Dar AlTeb subfertility centre, Cairo, Egypt

REFERENCES:
- [Background] Handyside AH, Kontogianni EH, Hardy K, Winston RM. Pregnancies from biopsied human preimplantation embryos sexed by Y-specific DNA amplification. Nature. 1990 Apr 19;344(6268):768-70. doi: 10.1038/344768a0. PMID 2330030
- [Background] Harton GL, De Rycke M, Fiorentino F, Moutou C, SenGupta S, Traeger-Synodinos J, Harper JC; European Society for Human Reproduction and Embryology (ESHRE) PGD Consortium. ESHRE PGD consortium best practice guidelines for amplification-based PGD. Hum Reprod. 2011 Jan;26(1):33-40. doi: 10.1093/humrep/deq231. Epub 2010 Oct 21. PMID 20966462
- [Background] Klitzman R, Zolovska B, Folberth W, Sauer MV, Chung W, Appelbaum P. Preimplantation genetic diagnosis on in vitro fertilization clinic websites: presentations of risks, benefits and other information. Fertil Steril. 2009 Oct;92(4):1276-1283. doi: 10.1016/j.fertnstert.2008.07.1772. Epub 2008 Sep 30. PMID 18829009
- [Background] Haapaniemi Kouru K, Malmgren H, Nordenskjold M, Fridstrom M, Csemiczky G, Blennow E. One-cell biopsy significantly improves the outcome of preimplantation genetic diagnosis (PGD) treatment: retrospective analysis of 569 PGD cycles at the Stockholm PGD centre. Hum Reprod. 2012 Sep;27(9):2843-9. doi: 10.1093/humrep/des235. Epub 2012 Jun 26. PMID 22736325
- [Background] Olivius C, Friden B, Borg G, Bergh C. Why do couples discontinue in vitro fertilization treatment? A cohort study. Fertil Steril. 2004 Feb;81(2):258-61. doi: 10.1016/j.fertnstert.2003.06.029. PMID 14967352
- [Background] Sills ES, Palermo GD. Preimplantation genetic diagnosis for elective sex selection, the IVF market economy, and the child--another long day's journey into night? J Assist Reprod Genet. 2002 Sep;19(9):433-7. doi: 10.1023/a:1016819908612. PMID 12408539
- [Background] Ehrich K, Williams C, Farsides B, Sandall J, Scott R. Choosing embryos: ethical complexity and relational autonomy in staff accounts of PGD. Sociol Health Illn. 2007 Nov;29(7):1091-106. doi: 10.1111/j.1467-9566.2007.01021.x. PMID 18092985
- [Background] Inzunza J, Iwarsson E, Fridstrom M, Rosenlund B, Sjoblom P, Hillensjo T, Blennow E, Jones B, Nordenskjold M, Ahrlund-Richter L. Application of single-needle blastomere biopsy in human preimplantation genetic diagnosis. Prenat Diagn. 1998 Dec;18(13):1381-8. doi: 10.1002/(sici)1097-0223(199812)18:133.0.co;2-n. PMID 9949438